CLINICAL TRIAL: NCT02717559
Title: Multicenter Orthopaedic Outcomes Network (MOON) ACL Reconstruction (ACLR): 10 Year Onsite Follow-up
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: The Cleveland Clinic (Other); Ohio State University (Other); Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Kurt P. Spindler, Adjoint Professor, Vanderbilt University Medical Center
Other Study IDs: 160049
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases
Keywords: Anterior cruciate ligament / injuries; Anterior cruciate ligament / surgery; knee injuries / surgery; outcomes research; prospective studies; osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Anterior Cruciate Ligament Injuries; Knee Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study the investigators will examine patients who have undergone unilateral ACL reconstruction surgery to determine which structural and functional characteristics of the knee two and ten years post reconstruction surgery, aspects of the original injury and repair, and patient characteristics are risk factors for osteoarthritis after ACL reconstruction surgery.

DETAILED DESCRIPTION:
The purpose of this study is to identify risk factors for signs and symptoms of osteoarthritis two and ten year post ACL reconstruction from information available at the time of surgery. Hypothesis: Smoking status, older age, higher BMI, increased severity of cartilage injuries, increased meniscal resection, revision surgery, and incidence of additional arthroscopic procedures will result in more symptoms and signs of osteoarthritis at 10-year follow-up.

Primary outcome measures will be the joint space width measured on weight-bearing radiographs, as well as the pain subscale of the Knee Injury and Osteoarthritis Score (KOOS).

Secondary outcome measures will include the knee related quality of life subscale of the Knee Injury and Osteoarthritis Score (KOOS).

ELIGIBILITY:
Inclusion Criteria:

* Had primary unilateral ACL reconstruction performed by Dr. Kurt Spindler (Vanderbilt University), Dr. Christopher Kaeding (The Ohio State University), Dr. Rick Parker (Cleveland Clinic), Dr. Jack Andrish (Cleveland Clinic), Dr. Rick Wright (Washington University, St. Louis), or Dr. Matthew Matava (Washington University, St. Louis).
* Participated in the 2 yr onsite visit

Exclusion Criteria:

* Unable to be consented
* Unable to participate for health reasons
* History of intra-articular knee infection
* History of total knee arthroplasty on either knee

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants enrolled in the Multicenter Orthopaedic Outcomes Network cohort by one of study site surgeons and meeting eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2016-03; Primary Completion 2025-12 (Actual); Study Completion 2025-12 (Actual)

PRIMARY OUTCOMES:
Joint space width measured on weight-bearing radiographs | 10 years after ACL reconstruction surgery
Pain subscale of the Knee Injury and Osteoarthritis Score (KOOS). | 10 years after ACL reconstruction surgery

SECONDARY OUTCOMES:
Knee related quality of life subscale of the Knee Injury and Osteoarthritis Score (KOOS) | 10 years after ACL reconstruction surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kurt P Spindler, MD, Principal Investigator — Vanderbilt University / The Cleveland Clinic Foundation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] MOON Group; Everhart JS, Jones MH, Yalcin S, Reinke EK, Huston LJ, Andrish JT, Cox CL, Flanigan DC, Kaeding CC, Magnussen RA, Obuchowski N, Parker RD, Pedroza AD, Sanders RA, Winalski CS, Spindler KP. The Clinical Radiographic Incidence of Posttraumatic Osteoarthritis 10 Years After Anterior Cruciate Ligament Reconstruction: Data From the MOON Nested Cohort. Am J Sports Med. 2021 Apr;49(5):1251-1261. doi: 10.1177/0363546521995182. PMID 33793363